CLINICAL TRIAL: NCT01633138
Title: Pilot Study of Performance-based Reinforcement to Enhance Cognitive Remediation Therapy for Substance Users
Brief Title: Performance-based Reinforcement to Enhance Cognitive Remediation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205010253; P50DA009241 (NIH)
Record Dates: First submitted 2012-06-27; First posted 2012-07-04 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Substance-Related Disorders; Mental Disorders
Keywords: cognitive remediation therapy; substance abuse treatment
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-S (Active Comparator): Cognitive Remediation Therapy - Standard
  Interventions: Behavioral: Cognitive Remediation Therapy - Standard
- CRT-CM (Experimental): Cognitive Remediation Therapy plus Contingency Management
  Interventions: Behavioral: Cognitive Remediation Therapy plus Contingency Management

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy - Standard — Computerized cognitive remediation therapy provided three times per week for four weeks
  Arms: CRT-S
Behavioral: Cognitive Remediation Therapy plus Contingency Management — Standard cognitive remediation therapy plus monetary incentives based on performance provided three times per week for four weeks.
  Arms: CRT-CM

SUMMARY:
The purpose of this study is to investigate whether monetary reinforcement for performance will enhance the effects of cognitive remediation therapy for substance users seeking treatment at an outpatient facility.

DETAILED DESCRIPTION:
Forty individuals seeking treatment for an alcohol or cocaine use disorder at the Substance Abuse Treatment Unit (SATU) will be randomized to receive cognitive remediation therapy with or without additional compensation based on performance. Participants will use the computerized cognitive remediation program (PSSCogRehab 2012) three times per week for four weeks. The primary outcome measure will be an improved performance on the computerized tasks, with secondary outcomes of changes in cognitive functioning (e.g., attention, concentration, memory) as measured by neuropsychological tests between baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* Primary Alcohol and/or Cocaine Abuse/Dependence Diagnosis
* Abstinence from all drugs/alcohol for 30 days
* Mild cognitive impairment
* Sufficiently stable and plan to commit to 4 weeks of outpatient treatment
* Fluent in English and 6th grade reading ability

Exclusion Criteria:

* Severe cognitive impairment indicative of dementia
* Untreated bipolar or psychotic disorder
* Have current legal case pending such that incarceration during 4-week study is likely

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement in performance scores on computerized cognitive remediation tasks | 4 weeks
  Performance scores on various computerized cognitive remediation tasks will be measured repeatedly during the 4 week study. These scores include "time to completion", "number of errors", "number of words correctly recalled", and "percentage of task completed"

SECONDARY OUTCOMES:
Improved cognitive function on neuropsychological tests | 4 weeks
  Change in cognitive function between baseline and post-treatment will be measured by performance on neuropsychological tests, such as Trail Making Test A & B, Wisconsin Card Sort Test, Digit Symbol Test from WAIS-IV, and the Continuous Performance Test-II (CPT-II).

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Kiluk, PhD, Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Unit, New Haven, Connecticut, United States